CLINICAL TRIAL: NCT01087333
Title: A Study of Hairy Cell and Other Leukemias With a Focus on Recombinant Immunotoxins for Cancer Treatment
Brief Title: Collection of Human Samples to Study Hairy Cell and Other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100066; 10-C-0066
Record Dates: First submitted 2010-03-13; First posted 2010-03-16 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-10-16

CONDITIONS: Hairy Cell Leukemia (HCL); Chronic Lymphocytic Leukemia (CLL); Non-Hodgkins Lymphoma (NHL); Cutaneous T Cell Lymphoma (CTCL); Adult T Cell Lymphoma (ATL)
Keywords: Cytotoxicity Assay; Neutralizing Antibodies; Apheresis; Flow Cytometry; Hemolytic Uremic Syndrome (HUS); Natural History
MeSH Terms: conditions — Leukemia, Hairy Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hemolytic-Uremic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with hematologic malignancies or solid tumors.
- 2: Normal Donors who are defined as individuals without a diagnosis of or history of any cancer.

SUMMARY:
Background:

- Researchers who are studying hairy cell leukemia, and how the disease compares with other disorders, are interested in obtaining additional samples from leukemia patients and healthy volunteers. The investigators are particularly interested in samples from individuals who have diseases that can be treated with a new type of drug called immunotoxin, in which an antibody carrying a toxin binds to a cancer cell and allows the toxin to kill the cell.

Objectives:

- To collect a variety of clinical samples, including blood, urine, lymph samples, and other tissues, in order to study the samples and develop new treatments for leukemia.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with leukemia or other kinds of blood and lymphatic system cancers, or who are healthy volunteers.

Design:

* Individuals who have leukemia will be asked to provide blood, bone marrow, urine, and tumor tissue samples as requested by the researchers. Healthy volunteers will provide only blood and urine samples.
* No treatment will be given as part of this protocol.

DETAILED DESCRIPTION:
Background

* Hairy cell leukemia (HCL) is highly responsive to but not curable by standard chemotherapy, and also responds well to investigational agents called recombinant immunotoxins which have been developed by the Laboratory of Molecular Biology (LMB).
* HCL variants often resemble classic HCL but are more aggressive and less responsive to treatments, such as HCLv and IGHV4-34+ HCL that are immunophenotypically indistinguishable from classic HCL and highly aggressive and resistant like HCLv.
* The investigators on this protocol are studying molecular and clinical aspects of HCL, and how they compare to normal or to other disorders, including other hematologic malignancies and solid tumors.
* The LMB are also studying agents for HCL/HCLv, including recombinant immunotoxins developed in the LMB. Specific targets and agents include BL22 and a high affinity variant, HA22 or Moxetumomab Pasudotox (Moxe), targeting CD22, LMB-2, targeting CD25, and SS1P, targeting Mesothelin as well as single agents and combinations of purine analogs (e.g., cladribine, pentostatin, and bendamustine), anti-CD20 monoclonal antibodies (e.g., rituximab), and small molecule inhibitors (e.g., BRAF V600E inhibitors dabrafenib and encorafenib, MEK inhibitors trametinib and binimetinib, and Bruton s tyrosine kinase (BTK) inhibitor ibrutinib).
* Longitudinal evaluation of HCL is needed as a basis to identify more effective treatments.

Objective

-To allow the collection and analysis of a variety of samples, including blood, tumor and other tissues from individuals with and without cancer to better understand the disease processes which are being studied, particularly hairy cell leukemia, or to determine eligibility and/or optimal timing for clinical testing

Eligibility

* Greater than or equal to 18 years of age
* Diagnosis of a hematologic malignancy or solid tumor; or normal donors (i.e., individuals without a known malignancy).

Design

* Collection of data and samples for research, including blood, tumor, and other tissues from participants and normal volunteers.
* Samples may be obtained prior to/after treatment, during disease assessments, and at the time of response/relapse. This protocol does not involve treatment, although participants may receive treatment as standard of care or as part of another research protocol during participation.
* Samples can be obtained at NIH or at local providers (and sent to NIH).
* Systematic follow-up of participants with HCL, in particular those who have completed prior treatment.
* We anticipate accruing 1263 participants on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants

* 18 years of age and older
* Desire of the individual to submit data and samples for research
* Ability to understand and the willingness to sign a written informed consent document.

Individuals with cancer

-Participants may have a diagnosis of hematologic malignancy or solid tumor. These participants would not be excluded if they were in long-term complete remission.

Normal donors (Individuals without cancer)

-Individuals must not have a current or prior diagnosis of a hematologic malignancy or solid tumor.

EXCLUSION CRITERIA:

All participants

-Known pregnancy at enrollment. NOTE: A pregnancy test will be required in individuals on study prior to any procedure done for research purposes that is greater than minimal risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary clinical population; normal donors
Sampling Method: Non-Probability Sample
Enrollment: 1263 (Estimated)
Dates: Start 2010-03-02 (Actual)

PRIMARY OUTCOMES:
Tissue Acquisition | 4 weeks
  Collection of a variety of clinical samples, including blood, urine, lymphapheresis samples, and other tissues and associated data

SECONDARY OUTCOMES:
HCL follow-up | about every 2 years
  Assess long-term treatment complications and disease outcomes in participants with HCL/HCLv

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Kreitman RJ, James L, Feurtado J, Eager H, Sierra Ortiz O, Gould M, Shpilman I, Zhou H, Burbelo PD, Cohen JI, Wang HW, Yuan CM, Arons E. COVID-19 vaccination in patients with classic and variant hairy cell leukemia. Blood Neoplasia. 2024 Aug 28;1(4):100035. doi: 10.1016/j.bneo.2024.100035. eCollection 2024 Dec. PMID 40552139
- [Derived] Arons E, Tai CH, Suraj J, Liu Y, Day CP, Raffeld M, Xi L, Zhou H, Gould M, Shpilman I, Oakes CC, Bhat S, Grever M, Jones D, Rogers K, Wang HW, Yuan CM, Sahinalp C, Kreitman RJ. Non-V600E BRAF mutations and treatment for hairy cell leukemia. Blood. 2025 Apr 24;145(17):1957-1961. doi: 10.1182/blood.2024026894. PMID 39719040
- [Derived] Arons E, Henry K, Haas C, Gould M, Tsintolas J, Mauter J, Zhou H, Burbelo PD, Cohen JI, Kreitman RJ. Characterization of B-cell receptor clonality and immunoglobulin gene usage at multiple time points during active SARS-CoV-2 infection. J Med Virol. 2023 Oct;95(10):e29179. doi: 10.1002/jmv.29179. PMID 37877800
- [Derived] Kreitman RJ, Yu T, James L, Feurtado J, Eager H, Ortiz OS, Gould M, Mauter J, Zhou H, Burbelo PD, Cohen JI, Wang HW, Yuan CM, Arons E. COVID-19 in patients with classic and variant hairy cell leukemia. Blood Adv. 2023 Dec 12;7(23):7161-7168. doi: 10.1182/bloodadvances.2023011147. PMID 37729613
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-C-0066.html